CLINICAL TRIAL: NCT05975164
Title: A Retrospective Real-world Study of Orelabrutinib in the Treatment of Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: the Real World Study of Orelabrutinib in the Treatment of CLL/SLL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Chunyan Ji, Prof., Shandong University
Other Study IDs: Orelabrutinib in real world
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: CLL/SLL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a Multicenter, Retrospective Real-world Study of Orelabrutinib in the Treatment of Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma in China

DETAILED DESCRIPTION:
Orelabrutinib is a novel BTK inhibitor with high selectivity and has been approved in China for relapsed/refractory CLL/SLL,, The purpose of this study is to describe the effectiveness and safety of orelabrutinib of chronic lymphocytic leukemia (CLL) in real world.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Patients with a definite diagnosis of CLL/SLL
3. Prior or current use of orelabrutinib for ≥3 months
4. At least one follow-up was recorded during orelabrutinib treatment

Exclusion Criteria:

1.Patients who received orelabrutinib in a prospective clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received orelabrutinib in real world
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-25 (Estimated); Primary Completion 2023-12-10 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | up to two years
  The ORR will be calculated as the proportion of participants who achieve either complete response (CR), partial response (PR) or partial response with lymphocytosis, as assessed by the participating physician.

SECONDARY OUTCOMES:
Time to Next Therapy (TTNT) | up to two years
  The TTNT will be calculated as the difference betweenorelabrutinib initiation date and initiation date of the first next therapy for CLL
Progression Free Survival (PFS) | up to two years
  PFS is defined as the duration from date of orelabrutinib initiation to date of disease progression (PD [according to the physician's evaluation]) or death from any cause
response rate of Hematologic Parameters | up to two years
  the proportion of participants who had abnormal baseline hemoglobin, or platelet, or lymphocyte counts returned to normal levels or had ≥50% increases in hemoglobin and platelets or ≥50% decreases in lymphocyte counts
safety | up to two years
  Percentage of Participants with Adverse Events (AEs), Serious Adverse Events (SAEs) and Special Situations

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Ji, Dr., Principal Investigator — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: Undecided